CLINICAL TRIAL: NCT03364790
Title: Correlation Between the Lower Extremities and Lumbar Degenerative Diseases of the Elderly and Formulation on Treatment Principles
Brief Title: Correlation Between the Lower Extremities and Lumbar Degenerative Diseases of the Elderly
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Liu Haiying, Department of spinal surgery, Peking University People's Hospital
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: Lumbar and Knee
Record Dates: First submitted 2017-11-25; First posted 2017-12-07 (Actual); Last update posted 2017-12-07 (Actual); Status verified 2017-12

CONDITIONS: Lumbar Osteoarthritis
Keywords: knee - spine syndrome; PLIF; TKA; sagittal parameters; neuroelectrophysiology
MeSH Terms: conditions — Osteoarthritis, Spine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- group1 (Experimental): participant with posterior lumbar interbody fusion(PLIF or PLF)
  Interventions: Procedure: PLIF
- group2 (Experimental): participant with total knee arthroplasty (TKA)
  Interventions: Procedure: TKA
- group3 (Experimental): participant with PLIF and TKA on one stage
  Interventions: Procedure: PLIF; Procedure: TKA
- group4 (No Intervention): participant without operation

INTERVENTIONS:
Procedure: PLIF — Randomly include the 30 participants diagnosed LSS and knee arthritis or limited by knee extension greater than 10 °who need to be operated and then performed PLIF or PLF; include anothr ones of 30 need to be with the implementation of TKA;and another group with the same diagnosis will be underwent both of surgeries in one stage.
  Arms: group1; group3
Procedure: TKA — Randomly include the 30 participants diagnosed LSS and knee arthritis or limited by knee extension greater than 10 °who need to be operated and then performed PLIF or PLF; include anothr ones of 30 need to be with the implementation of TKA;and another group with the same diagnosis will be underwent both of surgeries in one stage.
  Arms: group2; group3

SUMMARY:
The study has before mentioned the concept of "knee - spine syndrome" domestically, on the basement of which, the new study intends to perform another further study on the relationship between lumbar and lower extremity degenerative diseases.

DETAILED DESCRIPTION:
A prosepective, single-center, factorial design, randomized study will be performed. In this study, the 120 participants with degenerative lumbar and knees disease coped with the standard were included, then were assigned into 4 groups randomly. The patients in 3 operation groups were treated with posterior lumbar interbody fusion(PLIF or PLF) or total knee arthroplasty (TKA) or both of them in one stage respectively and the forth group with no surgery. The comparison between observation and operation group and the difference on self-control pre-and post-operatively in operation group within 6 months were measured and valuated. The result will be formed by the correlation and causal relationship on sagittal parameters on photograph, biomechanics, neuroelectrophysiology and molecular biology and the conclusions drawn by the use of modern medical basic research methods will formulate the treatment principles on it.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed LSS need to be underwent PLIF or PLF
2. and Patients who need surgery and are limited by knee extension greater than 10 °
3. ineffective conservative treatment for 6 months
4. patients have never relevant surgery before
5. Participants will be volunteered randomly assigned to surgery group and observation group.

Exclusion Criteria:

1. People have had similar lumbar or knee surgery
2. patients with lumbar or knee joint tumor or congenital malformation
3. there are contraindications of surgery such as infections and serious illness.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2020-12-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Body angle | 6 months
  Body angle is defined an angle of the shoulder and femoral trochanter connection and the greater trochanter and knee lateral condyle connection.

SECONDARY OUTCOMES:
Lumbar lordosis angle (LL) | 6 months
  Lumbar lordosis angle
Lumbar spinal area | 6 months
  measured by CT(GE light speed QX/i)
knee extension angle | 6 months
  The angle of knee extension the angle between the line connecting the greater trochanter of the femur and the lateral condyle of the femur and the line connecting the lateral condyle of the knee and the lateral condyle of the ankle.

CONTACTS AND LOCATIONS:
Overall Officials: Haiying Liu, Principal Investigator — Department of spinal surgery

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lin SI, Lin RM. Sensorimotor and balance function in older adults with lumbar nerve root compression. Clin Orthop Relat Res. 2002 Jan;(394):146-53. doi: 10.1097/00003086-200201000-00017. PMID 11795726
- [Background] Matsuyama Y, Hasegawa Y, Yoshihara H, Tsuji T, Sakai Y, Nakamura H, Kawakami N, Kanemura T, Yukawa Y, Ishiguro N. Hip-spine syndrome: total sagittal alignment of the spine and clinical symptoms in patients with bilateral congenital hip dislocation. Spine (Phila Pa 1976). 2004 Nov 1;29(21):2432-7. doi: 10.1097/01.brs.0000143671.67779.14. PMID 15507807
- [Background] Murata Y, Takahashi K, Yamagata M, Hanaoka E, Moriya H. The knee-spine syndrome. Association between lumbar lordosis and extension of the knee. J Bone Joint Surg Br. 2003 Jan;85(1):95-9. doi: 10.1302/0301-620x.85b1.13389. PMID 12585585